CLINICAL TRIAL: NCT07343388
Title: Evaluation of the Impact of Preoperative Anxiety on Postoperative Pain and Emergence Delirium in Patients Undergoing Pediatric Urogenital Surgery: A Prospective Observational Study
Brief Title: Relationship Between Preoperative Anxiety, Postoperative Pain, and Emergence Delirium in Pediatric Surgery
Status: Recruiting | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Collaborators: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, Gonul Sari, MD, Aydin Adnan Menderes University
Other Study IDs: GOA-155
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain; Preoperative Anxiety; Emergence Delirium in Pediatric Anesthesia; Urogenital Diseases
Keywords: preoperative anxiety; postoperative pain; Postoperative Complications; mYPAS; FLACC Scale; Aldrete Score; PAED Scale
MeSH Terms: conditions — Pain, Postoperative; Urogenital Diseases; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Urogenital Surgery Group
  Interventions: Other: Standardized Perioperative Management and Observational Assessment

INTERVENTIONS:
Other: Standardized Perioperative Management and Observational Assessment — All participants will undergo a standardized general anesthesia protocol for elective urogenital surgery (hypospadias repair, orchidopexy, or hydrocele surgery). The intervention includes:
  Preoperative Phase: Assessment of anxiety using the mYPAS scale before induction.
  Intraoperative Phase: Standardized induction and maintenance of anesthesia (e.g., inhalational anesthesia with sevoflurane).
  Postoperative Phase: Systematic observation in the Post-Anesthesia Care Unit (PACU) using Modified Aldrete, PAED, and FLACC scales at 0, 15, 30, 45, and 60 minutes. No experimental drugs or techniques will be administered; the study focuses on the observational correlation between preoperative anxiety and recovery outcomes."

SUMMARY:
The goal of this observational study is to learn if preoperative anxiety levels can predict the quality of early postoperative recovery, pain intensity, and the occurrence of emergence delirium in pediatric patients aged 2 to 7 years undergoing elective urogenital surgery, specifically hypospadias repair, orchidopexy, and hydrocele surgery.

The main questions it aims to answer are:

Does a higher level of preoperative anxiety lead to increased postoperative pain and a higher incidence of emergence delirium?

Is there a significant relationship between preoperative anxiety and the speed of physical recovery (discharge readiness) as measured by Aldrete scores?

Researchers will compare outcomes of patients with different levels of preoperative anxiety to see if higher anxiety results in poorer recovery profiles in the immediate postoperative period.

Participants will:

Be assessed for anxiety levels using the Modified Yale Preoperative Anxiety Scale (mYPAS) immediately before anesthesia induction.

Undergo a standardized anesthesia protocol for their elective urogenital procedure (hypospadias repair, orchidopexy, or hydrocele surgery).

Be monitored in the Post-Anesthesia Care Unit (PACU) at 0, 15, 30, 45, and 60 minutes after surgery to evaluate physical recovery (Modified Aldrete Score), delirium (PAED scale), and pain intensity (FLACC scale).

ELIGIBILITY:
Inclusion Criteria:

Male patients aged 2 to 7 years.

ASA (American Society of Anesthesiologists) physical status I or II.

Scheduled for elective urogenital surgery, specifically hypospadias repair, orchidopexy, or hydrocele surgery.

Scheduled to undergo general anesthesia for the procedure.

Patients with no history of neurological or psychiatric disorders.

Provision of written informed consent by the parents or legal guardians.

Exclusion Criteria:

* Patients outside the specified age range (younger than 2 or older than 7 years).

Female patients.

Patients undergoing emergency surgeries or non-urogenital/non-inguinal procedures.

Presence of a diagnosed cognitive impairment or developmental delay.

Parental or legal guardian refusal to provide informed consent.

Ages: 2 Years to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of pediatric patients aged 2 to 7 years who are scheduled for elective urogenital surgical procedures at a tertiary pediatric training and research hospital. The cohort specifically focuses on patients undergoing common inguinoscrotal surgeries, including hypospadias repair, orchidopexy, and hydrocele surgery, under standardized general anesthesia. Participants are selected from patients who meet the ASA I-II physical status criteria and have no underlying neurological or psychiatric conditions that could interfere with anxiety and delirium assessments.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Intensity | Postoperatively at 0, 15, 30, 45, and 60 minutes.
  Measured using the Face, Legs, Activity, Cry, Consolability (FLACC) scale. This behavioral scale assesses pain in children who cannot communicate verbally. Each of the five categories is scored from 0 to 2, resulting in a total score ranging from 0 to 10. Higher scores indicate increased pain intensity (0: Relaxed/Comfortable, 1-3: Mild discomfort, 4-6: Moderate pain, 7-10: Severe pain/discomfort).
Incidence and Severity of Emergence Delirium | Postoperatively at 0, 15, 30, 45, and 60 minutes.
  Measured using the Pediatric Anesthesia Emergence Delirium (PAED) scale. The scale consists of five items: eye contact, purposeful actions, awareness of surroundings, restlessness, and inconsolability. The total score ranges from 0 to 20, where higher scores indicate greater severity of delirium. A score of 10 or higher is considered clinically significant for the presence of emergence delirium.

SECONDARY OUTCOMES:
Postoperative Physical Recovery and Discharge Readiness | Postoperatively at 0, 15, 30, 45, and 60 minutes.
  Measured using the Modified Aldrete Score, which evaluates five criteria: activity, respiration, circulation, consciousness, and oxygen saturation. Each criterion is scored 0, 1, or 2. The total score ranges from 0 to 10. Higher scores indicate better physical recovery and greater readiness for discharge from the Post-Anesthesia Care Unit (PACU). A score of 9 or 10 is typically required for safe discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Behcet Uz Children's Hospital, Izmir, Konak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Topalel S, Orekici Temel G, Azizoglu M. Evaluation of Preoperative Anxiety in Turkish Paediatric Patients and Validity and Reliability of the Turkish Modified Yale Preoperative Anxiety Scale. Turk J Anaesthesiol Reanim. 2020 Dec;48(6):484-490. doi: 10.5152/TJAR.2020.116. Epub 2020 May 18. PMID 33313588